CLINICAL TRIAL: NCT01971645
Title: Dexamethasone as an Adjuvant to Ropivacaine for Femoral Nerve Blocks in Children Undergoing Knee Arthroscopy
Brief Title: Decadron as Adjuvant in Femoral Nerve Blocks in Knee Arthroscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Giorgio Veneziano, Assistant Clinical Professor, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB13-00610
Record Dates: First submitted 2013-10-22; First posted 2013-10-29 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Knee Injury
Keywords: Dexamethasone; Ropivacaine; Knee arthroscopy; Femoral nerve blocks; Peripheral nerve blocks; Adjuvant; Pediatrics
MeSH Terms: conditions — Knee Injuries | interventions — Dexamethasone; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group D (Experimental): Group D patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) with 0.1 mg/kg preservative-free dexamethasone (max. dose 4 mg) perineurally for their femoral block. Group D will also receive a gluteal intramuscular injection of saline of volume equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml).
  Interventions: Drug: Dexamethasone; Drug: Ropivacaine
- Group R (Placebo Comparator): Group R patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) combined with a volume of saline equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml) perineurally. Group R will also receive a gluteal intramuscular injection of saline of volume equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml).
  Interventions: Drug: Ropivacaine
- Group M (Active Comparator): Group M patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) combined with a volume of saline equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml) perineurally. Group M will also receive a gluteal intramuscular injection of 0.1 mg/kg preservative-free dexamethasone (max. dose 4 mg).
  Interventions: Drug: Dexamethasone; Drug: Ropivacaine

INTERVENTIONS:
Drug: Dexamethasone — Patients may receive 0.1 mg/kg preservative-free dexamethasone (max. dose 4 mg) either perineurally or intramuscularly.
  Arms: Group D; Group M
Drug: Ropivacaine — Patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) perineurally.

SUMMARY:
If preservative-free dexamethasone 0.1 mg/kg (max dose 4 mg) is added to ropivacaine 0.5% 2 mg/kg (max dose 100 mg), then post-PACU opioid consumption will be reduced by 33%.

DETAILED DESCRIPTION:
Following informed consent, patients will be randomized to one (1) of three (3) arms. Group D patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) with 0.1 mg/kg preservative-free dexamethasone (max. dose 4 mg) perineurally for their femoral block. Group D will also receive a gluteal intramuscular injection of saline of volume equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml). Group R patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) combined with a volume of saline equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml) perineurally. Group R will also receive a gluteal intramuscular injection of saline of volume equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml). Group M patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) combined with a volume of saline equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml) perineurally. Group M will also receive a gluteal intramuscular injection of 0.1 mg/kg preservative-free dexamethasone (max. dose 4 mg). The randomization will be blinded to the patient, surgery team, anesthesia team, recovery nurses, and clinical research nurses.

The remainder of the anesthetic care will remain the same per our usual routine for these cases. On arrival to the operating room:

1. Standard American Society of Anesthesiologists (ASA) monitors will be placed on the patient (ECG, pulse oximetry, non-invasive BP, thermistor).
2. A peripheral intravenous catheter will be placed while patient is inhaling 50% nitrous oxide.
3. Intravenous induction will be accomplished with midazolam 2 mg, propofol 2-3 mg/kg.
4. Once induction is complete, a laryngeal mask airway will be placed.
5. Maintenance of anesthesia will be provided with inhaled sevoflurane titration.
6. The femoral nerve block will be performed by one of the anesthesiologist co-investigators.
7. After completion of a pre-block time-out, the patient's groin on side of surgery will be prepped with chlorhexidine.
8. Using aseptic technique, a needle will be advanced under ultrasound guidance to the femoral nerve.
9. In addition to ultrasound, a nerve stimulator may be used at the anesthesiologist's discretion to help identify the femoral nerve.
10. After identification of the femoral nerve, the perineural study drug will be injected around the femoral nerve.
11. Using aseptic technique the intramuscular study drug will be injected into the gluteus muscle.
12. For intraoperative increases in heart rate or systolic blood pressure >20 % above levels immediately prior to incision, fentanyl will be given in 1 µg/kg increments every 5 minutes until below this threshold. (No acetaminophen, ketorolac, or IV dexamethasone will be given)
13. Once the patient arrives to PACU, dilaudid 5 µg/kg (max. dose 0.3 mg) every ten minutes may be given until patient VAS score is less than or equal to 4.
14. In the surgery unit, patients may receive one dose of hydrocodone-acetaminophen (7.5 mg/325 mg/15 ml) liquid suspension 0.1 mg/kg hydrocodone PO (max. dose 10mg hydrocodone) and then may receive dilaudid 5 µg/kg IV if pain persists above a VAS of 4 (max. dose 0.3 mg).
15. Patients will be discharged from the surgery unit with a prescription for hydrocodone-acetaminophen (7.5 mg/325 mg/15 ml) liquid suspension. The prescription will be for 0.1 mg/kg hydrocodone PO (max. dose 10 mg hydrocodone) every 4 hours as needed for all patients.
16. Patients will be sent home with a pain diary to record consumption of pain medication, when 1st dose of pain medications was taken, when sensory and motor blocks resolved and degree of motor block 24 and 48 hours according to the Bromage scale (Table 1). All adverse effects including nausea, vomiting, pruritus, excessive sedation will be asked to be recorded in the diary.
17. A clinical research nurse will collect information on opioid consumption on day of surgery (DOS) and intensity of motor block in PACU according to the Bromage scale.
18. On post-operative day 1 and 2 a clinical research nurse will call to collect information from the diary for analysis. If sensory or motor blockade persists on day 2, then the patient will be called on day 3. If neurologic symptoms persist after 72 hours, the patient will be asked to come to pre-operative clinic for a neurologic examination by an anesthesiologist. If neurological deficits are present on exam, the patient will be referred to a neurologist. Neurology will then determine if further testing is required. In addition, all patients will be contacted by telephone at 2 weeks after study initiation. If any new neurologic deficits are reported at this time, patients will be brought into the preoperative clinic and undergo the same evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Children older than 10, and younger than 19 years of age undergoing unilateral arthroscopic surgery of the knee
* American Society of Anesthesiologists (ASA) Status I or II
* Patient's parent/guardian willing and able to give consent
* Patient willing to give assent

Exclusion Criteria:

* Arthroscopic anterior cruciate ligament repair
* Systemic steroid use within the last 3 months
* Diabetes mellitus
* Females testing positive for pregnancy
* BMI > 98th percentile
* Positive pregnancy test
* Coagulopathy
* Renal or hepatic disease
* Pre-existing motor or sensory deficits in the lower extremities
* Predisposition for falls based on pre-existing sensory or motor deficits of the legs or inability to perform crutch training.
* Non-English speaking
* Systemic fungal infection
* Immunosuppressed patients

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Veneziano, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Veneziano G, Martin DP, Beltran R, Barry N, Tumin D, Burrier C, Klingele K, Bhalla T, Tobias JD. Dexamethasone as an Adjuvant to Femoral Nerve Block in Children and Adolescents Undergoing Knee Arthroscopy: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial. Reg Anesth Pain Med. 2018 May;43(4):438-444. doi: 10.1097/AAP.0000000000000739. PMID 29377866

RESULTS

PARTICIPANT FLOW:
Groups:
- Perineural Dexamethasone Group: Perineural group patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) with 0.1 mg/kg preservative-free dexamethasone (max. dose 4 mg) perineurally for their femoral block. Group D will also receive a gluteal intramuscular injection of saline of volume equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml).
  Dexamethasone: Patients may receive 0.1 mg/kg preservative-free dexamethasone (max. dose 4 mg) either perineurally or intramuscularly.
  Ropivacaine: Patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) perineurally.
- Ropivacaine Group: Ropivacaine group patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) combined with a volume of saline equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml) perineurally. Group R will also receive a gluteal intramuscular injection of saline of volume equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml).
  Ropivacaine: Patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) perineurally.
- Intramuscular Dexamethasone Group: Intramuscular group patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) combined with a volume of saline equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml) perineurally. Group M will also receive a gluteal intramuscular injection of 0.1 mg/kg preservative-free dexamethasone (max. dose 4 mg).
  Dexamethasone: Patients may receive 0.1 mg/kg preservative-free dexamethasone (max. dose 4 mg) either perineurally or intramuscularly.
  Ropivacaine: Patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) perineurally.
Period: Overall Study
Arm/Group | Perineural Dexamethasone Group | Ropivacaine Group | Intramuscular Dexamethasone Group
Started | 25 | 27 | 25
Completed | 23 | 27 | 23
Not Completed | 2 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Perineural Dexamethasone Group: Group D patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) with 0.1 mg/kg preservative-free dexamethasone (max. dose 4 mg) perineurally for their femoral block. Group D will also receive a gluteal intramuscular injection of saline of volume equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml).
  Dexamethasone: Patients may receive 0.1 mg/kg preservative-free dexamethasone (max. dose 4 mg) either perineurally or intramuscularly.
  Ropivacaine: Patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) perineurally.
- Ropivacaine Group: Group R patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) combined with a volume of saline equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml) perineurally. Group R will also receive a gluteal intramuscular injection of saline of volume equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml).
  Ropivacaine: Patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) perineurally.
- Intramuscular Dexamethasone Group: Group M patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) combined with a volume of saline equivalent to 0.1 mg/kg preservative-free dexamethasone (max. volume 0.4 ml) perineurally. Group M will also receive a gluteal intramuscular injection of 0.1 mg/kg preservative-free dexamethasone (max. dose 4 mg).
  Dexamethasone: Patients may receive 0.1 mg/kg preservative-free dexamethasone (max. dose 4 mg) either perineurally or intramuscularly.
  Ropivacaine: Patients will receive 2 mg/kg of 0.5% ropivacaine (max. dose 100 mg) perineurally.
- Total: Total of all reporting groups
Arm/Group | Perineural Dexamethasone Group | Ropivacaine Group | Intramuscular Dexamethasone Group | Total
Number analyzed (Participants) | 25 | 27 | 25 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 26 | 24 | 74
  Between 18 and 65 years | 1 | 1 | 1 | 3
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (2) | 14.6 (2) | 14.7 (2) | 14.8 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 16 | 41
  Male | 11 | 16 | 9 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 27 | 25 | 77

OUTCOME MEASURES:

1. Primary Outcome: Intra-operative and Post-operative Opioid Consumption
Description: Number of doses of narcotic pain medicine administered during surgery and up to 48 hours after discharge from surgery center.
Time Frame: Intra-operative and up to 48 hours post-discharge, an average of 48 hours
Measure: Median (Inter-Quartile Range); unit: doses
Arm/Group | Group D | Group R | Group M
Number analyzed (Participants) | 23 | 27 | 23
doses | 2 [1 to 4] | 2 [0 to 5] | 3 [0 to 6]

2. Secondary Outcome: Post-operative Pain Scores
Description: Visual Analogue Scale (VAS) pain scores (0 being no pain and 10 being worst pain) from arrival to post-anesthesia care unit (PACU) to 48 hours after discharge from surgery center.
Time Frame: Immediately post-operatively and up to 48 hours post-discharge, an average of 48 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group D | Group R | Group M
Number analyzed (Participants) | 23 | 27 | 23
units on a scale | 2 [0 to 4] | 2 [0 to 2] | 1 [0 to 3]

ADVERSE EVENTS:
Time Frame: From beginning of surgery until 2 weeks post-op, an average of 2 weeks.
Arm/Group | Group D | Group R | Group M
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 1/25 | 0/27 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group D (N=25) | Group R (N=27) | Group M (N=25)
emergence delerium (Injury, poisoning and procedural complications) | 1 | 0 | 0 — An abnormal mental state that develops as a result of anesthesia administration during the transition from unconsciousness to complete wakefulness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes